CLINICAL TRIAL: NCT00252369
Title: Instillation of Fibrin Glue After Induction of Local Conditions Using Infliximab, in the Treatment of Perianal Crohn's Disease.
Brief Title: Treatment of Perianal Crohn's Disease, Combining Medical and Surgical Treatment.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-05-3762-OZ-CTIL
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-04-24 (Estimated); Status verified 2009-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infliximab
Procedure: Instillation of fibrin glue

SUMMARY:
This study is aimed to assess the hypothesis that instillation of fibrin glue with the induction of local conditions using Infliximab, may be useful in the treatment of perianal Crohn's disease.

DETAILED DESCRIPTION:
Patients with perianal fistulae of Crohn's disease will be prospectively enrolled and receive 3 doses of Infliximab. If reduction of fistula associated discharge of at least 50% will be recorded, commercially available fibrin glue will be instilled into the fistula tract using standard surgical techniques. The patients will be followed for 6 months for fistula healing and complications.

ELIGIBILITY:
Inclusion Criteria:

* Perianal fistula of Crohn's dis

Exclusion Criteria:

* More then 2 fistulae perianal sepsis known contraindication to infliximab or glue

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Fistula healing

SECONDARY OUTCOMES:
Quality of life
Complications

CONTACTS AND LOCATIONS:
Overall Officials: Oded Zmora, MD, Principal Investigator — Sheba Medical Center
Locations (4):
- Israel (4):
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Assaf Harofe Medical Center, Zrifin